CLINICAL TRIAL: NCT03161288
Title: A Single and Multiple Ascending Dose, Placebo-Controlled, Double-Blind, Phase 1 Study of KY1005 in Healthy Volunteers
Brief Title: A Study of KY1005 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kymab Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY1005-CT01
Record Dates: First submitted 2017-05-11; First posted 2017-05-19 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Immune System Diseases
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohorts 1-3 (Experimental): Healthy volunteers will receive single rising doses of KY1005 or placebo
  Interventions: Drug: KY1005; Drug: Placebo
- Cohorts 4-8 (Experimental): Healthy volunteers will receive multiple rising doses of KY1005 or placebo
  Interventions: Drug: KY1005; Drug: Placebo

INTERVENTIONS:
Drug: KY1005 — A human anti-OX40 ligand monoclonal antibody
Drug: Placebo — Matched placebo

SUMMARY:
This is a single and multiple ascending dose, placebo-controlled, double-blind, Phase 1 study to evaluate the safety and tolerability of KY1005 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfil all of the following criteria for entry into the study.

1. Volunteer to participate in the clinical trial and provide signed informed consent.
2. Male, aged 18 to 45 years.
3. Subjects with a female spouse/partner of childbearing potential must agree to use effective birth control starting at screening and continuing throughout the clinical study period and for a period of up to 6 months after study completion.
4. Cohorts 4 to 8: previous immunisation with tetanus toxoid (TT) but not within 6 months prior to the screening visit as reported by the volunteer.
5. Cohorts 4 to 8: anti-TT immunoglobulin G (IgG) response > 0.1 IU/mL and ≤ 50 IU/mL at screening.

Exclusion Criteria:

Subjects fulfilling any of the following exclusion criteria are not eligible for entry into the study.

1. Experiencing a clinically significant, chronic or acute infection requiring treatment at screening or prior to first IMP administration.
2. A body weight of ≤ 60.0 kg or ≥ 120.0 kg.
3. A body mass index ≤ 18.0 or ≥ 30.0 kg/m2.
4. History of disease of the central nervous system, cardiovascular system, kidney, liver, digestive system, respiratory system or metabolic/endocrine system or suffered from other disease that in the opinion of the principal investigator (or medically qualified designee) may make participation unsafe for the subject or interfere with trial evaluations or otherwise considered clinically significant.
5. History of immunological abnormality (e.g., immune suppression, severe allergy or anaphylaxis) that in the opinion of the principal investigator (or medically qualified designee) may make participation unsafe for the subject or interfere with trial evaluations or otherwise considered clinically significant.
6. History of malignancy, or known current malignancy.
7. Leukocyte absolute value < 3.50 × 10^9/L or > 9.50 × 10^9/L, neutrophil absolute value < 1.8 × 10^9/L, platelet counts < 100 × 10^9/L, haemoglobin < 12.0 g/dL.
8. Taken part in other clinical trials within 3 months of screening for this study or > four trials in the year preceding the first IMP administration.
9. Donated or lost more than 500 mL of blood or plasma within 3 months of screening.
10. Prescription drug taken within 2 weeks of screening or likely to be taken during the trial.
11. Live immunisation within 3 months of screening or plans to receive such immunisation during the clinical trial or for a period of 6 months after the end of the trial.
12. Taking or likely to take over-the-counter medication, including herbal medicines, that in the opinion of the principal investigator (or medically qualified designee) may make participation unsafe for the subject or interfere with trial evaluations.
13. Hepatitis B surface antigen, Hepatitis C antibody, or Human Immunodeficiency Virus positive.
14. History of or current drug or substance abuse considered significant by the principal investigator (or medically qualified designee) including a positive urine drug screen.
15. Current smoker and/or regular user of other nicotine-containing products (e.g., patches).
16. Average consumption of more than 14 units of alcohol/week.
17. Clinically significant abnormal screening values in clinical (electrocardiograms (ECGs), vital signs, physical examination) and laboratory tests in the opinion of the principal investigator (or medically qualified designee).
18. Cannot communicate adequately or cannot commit to full participation in all trial procedures.
19. For Cohorts 4 to 8:

    1. Confirmed previous exposure to immunocyanins, such as keyhole limpet haemocyanin (KLH);
    2. Known allergy to thiomersal or other components of Tetanus vaccine or Immucothel®;
    3. History of schistosomiasis.
20. Any observation that, in the opinion of the principal investigator (or medically qualified designee) makes the subject unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male volunteers.
Enrollment: 64 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of all treatment-related adverse events | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
Changes in vital signs (as a measure of safety and tolerability) | Cohorts 1 to 3: from pre-first infusion up to day 113. Cohorts 4 to 8: from pre- first infusion up to day 92.
Changes in laboratory safety data (as a measure of safety and tolerability) | Cohorts 1 to 3: from pre-first infusion up to day 113. Cohorts 4 to 8: from pre-first infusion up to day 92.
Changes in anti-viral antibody levels and viral DNA (as a measure of safety and tolerability) | Cohorts 1 to 3: from pre-first infusion up to day 113. Cohorts 4 to 8: from pre-first infusion up to day 92.
Changes in acute cytokines (as a measure of safety and tolerability) | Cohorts 1 to 3: from pre-first infusion up to day 113. Cohorts 4 to 8: from pre-first infusion up to day 92.
Changes in electrocardiograms (as a measure of safety and tolerability) | Cohorts 1 to 3: from pre-first infusion up to day 113. Cohorts 4 to 8: from pre-first infusion up to day 92.

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) following the first, second and third infusions for each KY1005 dose/dosing group | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
Time to maximum observed serum concentration (tmax) following the first, second and third infusions for each KY1005 dose/dosing group | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
Trough concentrations (Cmin) following the first and second infusions and 28 days after the third infusion | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
Areas under the plasma concentration-time curves (AUC) | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
Clearance (CL) | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
Apparent volume of distribution during terminal phase (Vz) | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
Apparent volume of distribution at steady state (Vss) | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
Half-life (t½) | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.

OTHER OUTCOMES:
Serum anti-KY1005 antibody titres | Cohorts 1 to 3: up to day 113. Cohorts 4 to 8: up to day 92.
  Change in serum anti-KY1005 antibody titres from pre-infusion.
Immunophenotype and OX40/OX40L expression | Cohorts 1- 8: up to day 85.
  Changes in specific cell subsets and expression of OX40/OX40L on each subset (where evaluable).
Neo-antigen and recall antigen immunological responses (cohorts 4-8 only) | up to day 85
  Change in anti-tetanus toxoid immunoglobulin G (IgG) and immunoglobulin M (IgM) titres in serum and anti-Immucothel® IgG and IgM titres in serum.
Delayed Type Hypersensitivity response in the skin after intradermal injection of Immucothel® or saline measured by Antera 3D® camera image analysis (cohorts 4-8 only) | Day 85 and 87
  Change in skin colour a and haemoglobin level (concentration of redness per unit area relative to region of interest)
Delayed Type Hypersensitivity response in the skin after intradermal injection of Immucothel® or saline measured by LSCI photography (cohorts 4-8 only) | Day 85 and 87
  Change in basal flow and flare

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Burggraaf, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saghari M, Gal P, Gilbert S, Yateman M, Porter-Brown B, Brennan N, Quaratino S, Wilson R, Grievink HW, Klaassen ES, Bergmann KR, Burggraaf J, van Doorn MBA, Powell J, Moerland M, Rissmann R. OX40L Inhibition Suppresses KLH-driven Immune Responses in Healthy Volunteers: A Randomized Controlled Trial Demonstrating Proof-of-Pharmacology for KY1005. Clin Pharmacol Ther. 2022 May;111(5):1121-1132. doi: 10.1002/cpt.2539. Epub 2022 Mar 1. PMID 35092305